CLINICAL TRIAL: NCT01097460
Title: MM-111-02-12-02: A Phase 1 Study of MM-111 in Combination With Herceptin in Patients With Advanced, Refractory Her2 Amplified, Heregulin Positive Breast Cancer
Brief Title: MM-111 in Combination With Herceptin in Patients With Advanced Her2 Amplified, Heregulin Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-111-02-12-02
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Breast Neoplasms
Keywords: HER2/HER3; Bispecific Antibody; Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer; HER2 Positive Breast Cancer; Trastuzumab; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — MM-111; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MM-111 + Herceptin (Experimental): MM-111 will be combined with Herceptin
  Interventions: Drug: MM-111 + Herceptin

INTERVENTIONS:
Drug: MM-111 + Herceptin — For Phase 1: Dose escalation cohorts, MM-111 and Herceptin are administered weekly or bi-weekly via IV
  Other Names: Trastuzumab

SUMMARY:
This is an open-label Phase 1 trial of MM-111 in combination with Herceptin.

DETAILED DESCRIPTION:
Phase 1: Safety and tolerability of the MM-111 + Herceptin combination will be evaluated and the recommended Phase 2 dose will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced breast cancer that is amplified for HER2, based on archived tumor biopsy (IHC 2+ or greater)
* Patients must have histologically or cytologically confirmed advanced breast cancer that is heregulin positive based on fresh tumor tissue biopsy
* The patient's cancer must have recurred, progressed or not responded to standard chemotherapy or other standard treatment. Prior therapies may include but are not limited to Herceptin, Tykerb (lapatinib), anthracyclines, and taxanes
* Patients must be ≥ 18 years of age
* Patients or their legal representatives must be able to understand and sign an informed consent
* Patients may have measurable (per RECIST 1.1) or non-measurable tumor(s) (for Phase 1)
* Patients should have ECOG Performance Score (PS) 0, 1 or 2 (for Phase 1).
* Patients should have a life expectancy of at least 12 weeks
* Patients must have adequate bone marrow reserves
* Patients must have adequate hepatic function
* Patients must have adequate renal function
* Patients must be recovered from the effects of any prior surgery, radiotherapy or other antineoplastic therapy.
* Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of MM-111.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients with an active infection or with an unexplained fever > 38.5°C (101.3° F) during screening visits or on the first scheduled day of dosing.
* Patients with untreated and/or symptomatic metastatic CNS malignancies.
* Patients with known hypersensitivity to any of the components of MM-111 or who have had hypersensitivity reactions to fully human monoclonal antibodies, including Herceptin.
* Patients who have received other recent antitumor therapy including:

  * Treatment with Herceptin within the 28 days prior to the first scheduled day of dosing with MM-111
  * Investigational therapy administered within the 28 days prior to the first scheduled day of dosing MM-111 (Dosing in less than 28 days' since receiving investigational therapy is acceptable once a time interval equal to at least five half-lives of the investigational agent has passed.)
  * Any standard chemotherapy, Tykerb (lapatinib) or radiation within 14 days (and having passed the time of any actual or anticipated toxicities) prior to the first scheduled dose of MM-111
* Patients who have previously received MM-111
* Patients with NYHA Class III or IV congestive heart failure or LVEF < 50%
* Patients with a history of allogeneic transplant
* Patients with known HIV, hepatitis B or C (if patients have previously been treated for hepatitis C and have undetectable viral loads, they can be considered eligible for the trial)
* Patients with any other medical or psychological condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Higgins, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Indiana University (IUPUI), Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Huntsman Cancer Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- MM-111 + Herceptin: MM-111 will be combined with Herceptin
  MM-111 and Herceptin: For Phase 1: Dose escalation cohorts, MM-111 and Herceptin are administered weekly or bi-weekly via IV
Period: Overall Study
Arm/Group | MM-111 + Herceptin
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MM-111 + Herceptin
Number analyzed (Participants) | 16
Age, Continuous [Median (Standard Deviation); unit: years] | 54 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent AE's
Time Frame: 2 years
Population: Patients that received at least one dose
Measure: Number; unit: participants
Arm/Group | MM-111 + Herceptin
Number analyzed (Participants) | 16
participants | 16

2. Secondary Outcome: To Determine the Recommended Phase 2 Doses of MM-111 + Herceptin in Combination
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | MM-111 + Herceptin
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MM-111 + Herceptin (N=16)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
TRACHEAL OBSTRUCTION (Injury, poisoning and procedural complications) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MM-111 + Herceptin (N=16)
DIARRHOEA (Gastrointestinal disorders) | 7 (7)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
FATIGUE (General disorders) | 8 (8)
MUCOSAL INFLAMMATION (General disorders) | 2 (2)
OEDEMA (General disorders) | 2 (2)
PAIN (General disorders) | 2 (2)
CHILLS (General disorders) | 1 (1)
LOCALISED OEDEMA (General disorders) | 1 (1)
DYSPNOEA (Reproductive system and breast disorders) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 2 (2)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 4 (4)
DIZZINESS (Nervous system disorders) | 2 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2)
DYSARTHRIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4)
ANXIETY (Psychiatric disorders) | 3 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
ASPARATATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLOOD UREA INCREASED (Investigations) | 1 (1)
CARDIAC MURMUR (Investigations) | 1 (1)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TRACHEAL OBSTRUCTION (Injury, poisoning and procedural complications) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
HOT FLASH (Vascular disorders) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1)
SINUS OPERATION (Surgical and medical procedures) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other